CLINICAL TRIAL: NCT00749515
Title: Pilot Pharmacokinetic Study In Patients With Inadequate Response To Deferasirox (Exjade)
Brief Title: Pilot Study for Patients With Poor Response to Deferasirox
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Ellis Neufeld, Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07090349; NIH/NHLBI 1 K12 HL087164-01
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Transfusion-dependent Hemachromatosis; Thalassemia Major; Sickle Cell Disease
Keywords: Thalassemia; Iron; Chelation
MeSH Terms: conditions — beta-Thalassemia; Anemia, Sickle Cell; Thalassemia | interventions — Deferoxamine; Deferasirox; lidofenin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): All patients received the same interventions of deferoxamine challenge, deferasirox dose with pharmacokinetic monitoring and HIDA scan. Then we compared responses between patients who were known to be slow responders to deferasirox and those who were known to be rapid responders (chelated well).
  Interventions: Drug: Deferoxamine; Drug: Deferasirox; Radiation: HIDA

INTERVENTIONS:
Drug: Deferoxamine — After a 3-day washout period from all chelation, all patients have a 12 hour infusion of 50mg/kg of deferoxamine with urine collection and pre and post blood sampling to assess iron and Total Iron Binding Capacity (TIBC) by atomic absorption.
  Other Names: Desferal
Drug: Deferasirox — After a 3-day washout period from all chelation, patients had a desferal challenge which was followed by a single dose of deferasirox, 35mg/kg orally with blood sampling taken pre-deferasirox and at intervals for 24 hours after the dose.
  Other Names: Exjade; ICL670
Radiation: HIDA — All patients had a HIDA scan to assess physiologic liver clearance capacity.

SUMMARY:
This purpose of this study is to understand the differences between people who have a good response to deferasirox (exjade) compared to people who have a poor response to this medication when used for transfusion-dependent iron overload.

The hypothesis is that patients with poor responses have physiologic barriers to deferasirox that may include absorption, pharmacokinetics of drug metabolism, hepatic clearance and/or genetic factors.

DETAILED DESCRIPTION:
The purpose of this trial is to examine three potential mechanisms of inadequate response to Exjade® in patients with transfusion dependent iron overload including patients with thalassemia syndromes, sickle cell disease and bone marrow failure.

Hypothesis: Patients have physiologic barriers to adequately respond to deferasirox that may include absorption, pharmacokinetics of drug metabolism, hepatic clearance and/or genetic factors.

Study objectives Primary objective

* To evaluate three potential mechanisms for inadequate response to deferasirox in a small cohort of patients with hemoglobinopathies.
* Oral pharmacokinetics measured with Cmax and AUC following standard dose deferasirox.
* Hepatobiliary excretory function
* Accessibility of chelatable iron pool by deferoxamine challenge Secondary objective(s)
* To identify risk factors that can predict adequate response including demographics, disease status, presence and severity of liver disease, trough levels of deferasirox at outpatient visits and pharmacogenomics.
* To investigate usefulness of potential surrogate measures of response including serum deferasirox levels, Hepatobiliary Iminodiacetic Acid (HIDA)nuclear medicine scan to evaluate hepatic excretory function and urinary iron excretion by deferoxamine challenge.

This is an investigator-initiated, pilot-scale, open-label physiological assessment of patients who respond poorly to deferasirox compared with patients who respond well. We plan to study 2 groups of patients: a)10 patients who have demonstrated poor responses and b) 5 control patients with good responses as defined further in the protocol. The study has two parts.

Part I: Both groups of patients will have inpatient physiological assessments with a dose of 35mg/kg of deferasirox.

Part II: Inadequate responders eligible to continue on deferasirox will continue on a dose of 35 mg/kg for three months during which time serial pharmacokinetic levels will be studied. The control patients will resume their previous clinically appropriate dosing (likely less than 35 mg/kg) and for three months have serial pharmacokinetic levels drawn as well.

The study will begin with an outpatient screening visit when demographics and historical information as well as a physical examination will be obtained and reviewed for eligibility. At that visit patients will be able to sign informed consent. Shortly thereafter patients will be admitted to the GCRC at Children's Hospital Boston for part I of the study, a 2-3 day stay during which PK and nuclear medicine studies will be performed as well as the deferoxamine urinary iron excretion challenge. Patients who are eligible will continue on to part II of the study, and for 3 months and will be monitored for compliance, PK and ferritin changes on appropriate deferasirox doses.

ELIGIBILITY:
Part I: Inclusion criteria for Inadequate responders

* Male or female patients with transfusion dependent iron overload including patients with thalassemia syndromes, sickle cell disease and bone marrow failure.
* Patients currently on Desferal (desferrioxamine) therapy will require a one day wash out prior to the first dose of study drug.
* Dose of deferasirox: >30 mg/kg/day of deferasirox for at least 3 months
* No improvement or worsening of liver iron content (LIC) if this has been evaluated on deferasirox in the 3 months preceding the baseline studies.
* Age greater than 6 years
* Serum Ferritin: Ferritin >1500 ng/ml and rising over three month period while on deferasirox.
* Patients had to achieve 'failure' as described above previously and may or may not currently be on deferasirox and may currently be having adequate responses on doses greater than or equal to 35 mg/kg/day of deferasirox.
* Life expectancy ≥ 6 months
* Written informed consent by the patient or for pediatric patients consent of the patient's legal guardian. The definition of the term 'pediatric' for enrollment and study conduct will be in accordance with Children's Hospital IRB. Parents or the legal guardians will be fully informed by the investigator as to the requirements of the study. Pediatric patients themselves will be informed according to their capabilities in a language and in terms that they are able to understand. Written informed consent will be obtained from their legal guardian on the patient's behalf in accordance with national legislation. If capable, all patients should also personally sign their written informed consent.

Part I: Inclusion criteria for good responders:

* Male or female patients with transfusion dependent iron overload including patients with thalassemia syndromes, sickle cell disease and bone marrow failure.
* Patients currently on Desferal (desferrioxamine) therapy will require a one day wash out prior to the first dose of study drug.
* Serum ferritin less than or equal to 1000 ng/ml or declining over a 3 month period on a dose of less than 30 mg/kg of deferasirox.
* Age greater than 6 years
* Life expectancy ≥ 6 months
* Written informed consent by the patient or for pediatric patients consent of the patient's legal guardian. The definition of the term 'pediatric' for enrollment and study conduct will be in accordance with Children's Hospital IRB. Parents or the legal guardians will be fully informed by the investigator as to the requirements of the study. Pediatric patients themselves will be informed according to their capabilities in a language and in terms that they are able to understand. Written informed consent will be obtained from their legal guardian on the patient's behalf in accordance with national legislation. If capable, all patients should also personally sign their written informed consent.

Exclusion criteria for Part I:

* Pregnancy (as documented in required screening laboratory test) or breast feeding
* History of non-compliance to medical regimens or patients who are considered potentially unreliable and/or not cooperative
* Patients with transfusion requirements equal to or more frequent than every three weeks.
* AST or ALT > 400 U/L during screening
* Patients with uncontrolled systemic hypertension
* Severe cardiac insufficiency (NYHA III or IV), with uncontrolled and/or unstable cardiac or coronary artery disease not controlled by standard medical therapy
* Patients who received treatment with systemic investigational drug within the past 4 weeks or topical investigational drug within the past 7 days or are planning to receive other investigational drugs while participating in the study
* Allergy to deferoxamine
* Known contraindication to having a nuclear medicine study
* Any other condition which in the opinion of the investigator would prevent completion of the trial.
* Prior possible toxicity is not an exclusion criteria for Part I because patients require a chelating agent of which there are only two Patients who are found to be ineligible after screening procedures will have this documented on the screening log. No further data will be collected in the CRF for these patients.

Exclusion criteria for Part II:

* Patients with unacceptable toxicity to deferasirox such as renal failure or worsening cardiac function
* Patients who have failed to achieve negative iron balance at the maximum tolerated dose of deferasirox
* Patients who require an alternative chelator for specific reasons
* Patients who are currently enrolled on conflicting therapeutic trials
* Patients with serum ferritin less than 500 ng/ml at screening
* Any other condition which in the opinion of the investigator would prevent completion of the trial

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Chirnomas, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Chirnomas D, Smith AL, Braunstein J, Finkelstein Y, Pereira L, Bergmann AK, Grant FD, Paley C, Shannon M, Neufeld EJ. Deferasirox pharmacokinetics in patients with adequate versus inadequate response. Blood. 2009 Nov 5;114(19):4009-13. doi: 10.1182/blood-2009-05-222729. Epub 2009 Sep 1. PMID 19724055
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2008 and June 2008, 15 patients were recruited who had transfusional iron overload, and had been on deferasirox for at least 6 months at some point in their chelation history. Ten (10) patients were recruited as inadequate responders and 5 were recruited as control patients with adequate response to deferasirox therapy.
Groups:
- Inadequate Responders: Patients having a rising ferritin trend over 3 consecutive months, at least one higher than 1500ng/mL (1500 µg/L) or rising liver iron documented by biopsy or change in T2 or Ferriscan magnetic resonance imaging (MRI) and on a dose of more than 30img/kg per day of deferasirox.
- Adequate Responders (Control): Patients having a ferritin trend below 1000 ng/mL (1000 µg/L) or documented declining liver iron burden by MRI or biopsy and on a dose of 30img/kg per day or less of deferasirox.
Period: Overall Study
Arm/Group | Inadequate Responders | Adequate Responders (Control)
Started | 10 | 5
Completed | 10 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inadequate Responders | Adequate Responders (Control) | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 2 | 9
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve of Deferasirox After a Dose of 35 mg/kg
Description: Area Under the Curve (AUC) 0 to 24 hours post dose
Time Frame: 0, 1, 2, 4, 6, 8, 12, and 24 hours post dose
Measure: Mean (Standard Deviation); unit: micromole/liter*hour
Arm/Group | Inadequate Responders | Adequate Responders (Control)
Number analyzed (Participants) | 10 | 5
micromole/liter*hour | 479.59 (259.42) | 1123.11 (63.4)
Statistical Analysis 1: Comparison: Inadequate Responders vs Adequate Responders (Control); Test type: Other; p < .001, t-test, 2 sided

2. Primary Outcome: Half-Life of Deferasirox
Description: All patients received the same interventions of deferoxamine challenge, deferasirox dose with pharmacokinetic monitoring. Then we compared responses between patients who were known to be slow responders to deferasirox and those who were known to be rapid responders (chelated well).
  Deferoxamine: After a 3-day washout period from all chelation, all patients have a 12 hour infusion of 50mg/kg of deferoxamine with urine collection and pre and post blood sampling to assess iron and Total Iron Binding Capacity (TIBC) by atomic absorption.
Time Frame: 0, 1, 2, 4, 6, 8, 12, and 24 hours post dose.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Inadequate Responders | Adequate Responders (Control)
Number analyzed (Participants) | 10 | 5
hour | 6.08 (2.01) | 7.83 (2.95)
Statistical Analysis 1: Comparison: Inadequate Responders vs Adequate Responders (Control); Test type: Other; p = .275, t-test, 2 sided

3. Primary Outcome: Volume of Distribution/Bioavailability of Deferasirox After a Dose of 35 mg/kg
Description: Volume of distribution/bioavailability (Vd/F)
Time Frame: 0, 1, 2, 4, 6, 8, 12, and 24 hours post dose
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Inadequate Responders | Adequate Responders (Control)
Number analyzed (Participants) | 10 | 5
liter | 10.33 (7.42) | 6.5 (2.67)
Statistical Analysis 1: Comparison: Inadequate Responders vs Adequate Responders (Control); Test type: Other; p = .178, t-test, 2 sided

4. Primary Outcome: Volume of Distribution/Bioavailability of Deferasirox After a Dose of 35 mg/kg
Description: Volume of distribution/bioavailability (Vd/F), adjusted per kilogram body weight
Time Frame: 0, 1, 2, 4, 6, 8, 12, and 24 hours post dose
Measure: Mean (Standard Deviation); unit: liter/kilogram
Arm/Group | Inadequate Responders | Adequate Responders (Control)
Number analyzed (Participants) | 10 | 5
liter/kilogram | 0.32 (0.25) | 0.13 (0.05)
Statistical Analysis 1: Comparison: Inadequate Responders vs Adequate Responders (Control); Test type: Other; p = .062, t-test, 2 sided

5. Primary Outcome: Clearance/Bioavailability of Deferasirox in Patients With Poor Response to Deferasirox Compared to Patients With Good Response After a Dose of 35 mg/kg
Description: Clearance/bioavailability (CL/F)
Time Frame: 0, 1, 2, 4, 6, 8, 12, and 24 hours post dose.
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Inadequate Responders | Adequate Responders (Control)
Number analyzed (Participants) | 10 | 5
liter/hour | 1.30 (.18) | 0.61 (0.22)
Statistical Analysis 1: Comparison: Inadequate Responders vs Adequate Responders (Control); Test type: Other; p = .104, t-test, 2 sided

6. Secondary Outcome: Number of Participants With Polymorphisms in Genes Known to be, or Potentially Involved, in Deferasirox Disposition
Description: Polymorphisms in genes known to be, or potentially involved, in deferasirox disposition: UGT1a1 (including the Gilbert syndrome promoter polymorphism, (TA)nTAA),UGT1a3, BRCP/ABCG2, MRP2/ABCC2. These genes were chosen because deferasirox is primarily eliminated by glucuronidation and subsequent biliary excretion.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Inadequate Responders | Adequate Responders (Control)
Number analyzed (Participants) | 10 | 5
Participants
  UGT1a1 | 10 | 5
  UGT1a3 | 10 | 5
  BCRP/ABCG2 | 10 | 5
  MRP2/ABCC2 | 10 | 5

ADVERSE EVENTS:
Time Frame: Adverse event are reported for at least 28 days following the last dose of study drug.
Arm/Group | Inadequate Responders | Adequate Responders (Control)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 0/10 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No